CLINICAL TRIAL: NCT05587686
Title: Frequency of Respiratory Acidosis and Alkalosis in the Emergency and Intensive Care Department of the IUCPQ-UL. Potential Impact of the Use of the Application VentilO
Brief Title: Potential Impact of the Use of the Application VentilO
Status: Active, not recruiting | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal Investigator, Laval University
Other Study IDs: 22267
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intubated patient during their stay in the IUCPQ-UL emergency or intensive care department
  Interventions: Other: VentilO application

INTERVENTIONS:
Other: VentilO application — This educational application provides clinicians with combinations of tidal volume and respiratory rate based on gender, height, weight, body temperature and patient type. The algorithm used is based on published data regarding ventilatory requirements in different populations (i.e. from intubated patients for scheduled surgery to the most severe ICU patients) and anatomical and instrumental dead space.
  The objective of this application is to help implement personalized protective ventilation in intubated patients according to their characteristics.
  After patient data entry in the VentilO appllication we will compare the recommended settings (for mechanical ventilation) vs the real clinicial settings done by clinician after patient intubation.We will evaluated the potential effect of the VentilO recommendation on the first arterial (or capillary) blood gases compared to the real settings.

SUMMARY:
Mechanical ventilation is a vital support associated with the treatment of patients with acute respiratory failure and in other indications such as surgery under general anesthesia, coma or shock. Optimization of settings during mechanical ventilation and implementation of protective ventilation help to avoid ventilation-induced injury, ensure adequate oxygenation and maintain adequate carbon dioxide concentration to avoid respiratory acidosis or alkalosis.

Similarly, there is also no clear recommendation, to our knowledge, for the initial setting of the respiratory rate. Therefore, initial settings are not always adequate and in the literature the frequency of respiratory acidosis is very high, reaching about half of the patients receiving mechanical ventilation.

VentilO, is an application that is available on smart phones. This educational application provides clinicians with initial settings and optimization of these settings based on gender, height, weight, body temperature and patient type. The algorithm used is based on published data regarding ventilatory requirements in different populations and the anatomical and instrumental dead space of patients.

The purpose of our study is to:

1. Assess whether ventilatory settings after intubation are appropriate.
2. To compare the ventilatory adjustments made by clinicians with those proposed by the VentilO appalication.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> or = 18 years old)
* New endotracheal intubation

Exclusion Criteria:

* Absence of arterial (or capillary) gas within two hours of intubation
* Absence of patient sizes available throughout the medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated patients during their stay in the IUCPQ-UL emergency or intensive care department
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
acid-base abnormalities on arterial (or capillary) blood gases | on the first result available of arterial(or capillary) blood gases after intubation; 2 hours maximum post intubation
  evaluate the frequency of acid-base abnormalities, either acidosis or alkalosis, of respiratory or mixed origin on the first arterial gases after intubation.
  Respiratory acidosis is defined as a pH < 7.35 with a PaCO2 > 45 mmHg, and respiratory alkalosis as a pH > 7.45 with a PaCO2 < 35 mmHg)
Improvement acid-base abnormalities with the VentilO application | on the first result available of arterial(or capillary) blood gases after intubation; 2 hours maximum post intubation
  * In case of respiratory acidosis: minute ventilation proposed by VentilO > set minute ventilation;
  * In case of respiratory alkalosis: proposed minute ventilation by VentilO < set minute ventilation
Impairement acid-base abnormalities with the VentilO application | on the first result available of arterial(or capillary) blood gases after intubation; 2 hours maximum post intubation
  * In case of respiratory acidosis: proposed minute ventilation by VentilO < set minute ventilation
  * In case of respiratory alkalosis: minute ventilation proposed by VentilO > set minute ventilation

SECONDARY OUTCOMES:
Occurence of optimal arterial (or capillary) blood gases result | on the first result available of arterial(or capillary) blood gases after intubation; 2 hours maximum post intubation
  An optimal arterial (or capillary) blood gases as defined by a pH between 7.35 and 7.45 with a PaCO2 between 36 and 45 mmHg
Severity of unbalance of arterial (or capillary) blood gases result | on the first result available of arterial(or capillary) blood gases after intubation; 2 hours maximum post intubation
  For acid-base abnormalities, they will be evaluated according to their level of severity: the frequency of moderate (pH between 7.30 and 7.34) and severe (pH < 7.30) acidoses, and the frequency of moderate (pH between 7.46 and 7.50) and severe (pH > 7.50) alkaloses.
  The frequency of moderate (PaCO2 between 46 and 50 mmHg) and severe (PaCO2 > 50 mmHg) hypercapnia, and the frequency of moderate (PaCO2 between 31 and 35 mmHg) and severe (PaCO2 < 31 mmHg) hypocapnia
hemodynamic instabilities | Between Hour0 to Hour1 after intubation
  arterial hypotension requiring vascular filling > 1000 ml and/or use of vasopressors or inotropes such as levophed or adrenaline at > 0.05 mcg/kg/min)
ICU length of stay | up to 90 days. ICU stay - ICU admission through ICU discharge or until death if occured
  ICU length of stay - ICU admission through ICU discharge
Hospital length of stay | up to 90 days. ICU stay - Emergency department admission through hospital discharge or until death if occured
  Hospital length of stay - Emergency department admission through hospital discharge
ICU mortality | up to 90 days. ICU admission through until death if occured
  Occurence of death during ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec, Canada